CLINICAL TRIAL: NCT06344208
Title: Predicting Toxicity in Elderly Patients With Head and Neck Cancer: Validating a Disease-oriented Toxicity Predictive Tool and Integrating it With Available Screening Tools for Better Outcomes
Brief Title: Predicting Toxicity in Elderly Patients With Head and Neck Cancer
Acronym: PREtoxEL
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1647
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Predicting toxicity in elderly patients with head and neck cancer:

validating a disease-oriented toxicity predictive tool and integrating it with avail-able screening tools for better outcomes.

DETAILED DESCRIPTION:
We aim to analyze clinical and biochemical variables to prospectively create and validate an independ-ent predictive score to identify the probability of G3-5 toxicity in HNC elderly patients candidated to a curative treatment with radiation treatment +/- systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 70 years
* Histological diagnosis of squamous cell or undifferentiated HNC in stage III-IV AJCC ed VIII (si-nonasal, nasopharynx, oral cavity, oropharynx, unknown primary with HPV pos, larynx and hy-popharynx) and candidated to curative non surgical treatment (radiotherapy alone, Chemora-diation with platinum salts; radiation+cetuximab)
* Evaluable disease accordingly to RECIST criteria 1.1
* Willing of sign a written informed consent
* Adequate organ function

Exclusion Criteria:

Patient with cancer in other sites than HN < than 2 years except for prostate cancer cT1-2, Gleason 3+3, NIMBC, initial Non Melanoma Skin Cancer, in situ cervical cancer)

* PS ECOG 3-4
* Patients who received systemic treatments in the past for other primary tumors

Ages: 70 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 300 pts from the outpa-tients oncology practice previously discussed at multisciplinary meeting (MD) All the patients with age ≥ 70 years old, diagnosed with HNC candidated to a curative treatment with radiotherapy +/- systemic therapy (chemotherapy or cetuximab) will be evaluated.
Sampling Method: Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Predicting toxicity in elderly patients with head and neck cancer | 2 years
  validating a disease-oriented toxicity predictive tool and integrating it with avail-able screening tools for better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute of Oncology, Milan, Italy